CLINICAL TRIAL: NCT00845962
Title: Spinal Anesthesia With Bupivacaine or 2-chloroprocaine for Outpatient Elective Surgery: a Prospective, Randomized, Double-blind Comparison.
Brief Title: A Comparison of Bupivacaine and 2-chloroprocaine for Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Jean-Denis Roy / MD Anesthesiologist, Centre hospitalier de l'université de Montréal (CHUM) / University of Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD07.007; 118046
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2009-07

CONDITIONS: Spinal Anesthesia
Keywords: bupivacaine; chloroprocaine; spinal; anesthesia; elective surgery; ambulatory surgery
MeSH Terms: interventions — chloroprocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chloroprocaine (Active Comparator)
  Interventions: Drug: chloroprocaine
- Bupivacaine (Active Comparator)
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: chloroprocaine — spinal administration of chloroprocaine 2%, 40 mg (2 mL)
  Other Names: Nesacaine
  Arms: Chloroprocaine
Drug: bupivacaine — spinal administration of bupivacaine 0,75% 7,5 mg (1 mL)
  Other Names: Marcaine
  Arms: Bupivacaine

SUMMARY:
The purpose of this study is to compare the efficacity and the readiness for discharge between two local anesthetics, bupivacaine and 2-chloroprocaine, used for spinal anesthesia.

DETAILED DESCRIPTION:
Many surgeries are performed under spinal anesthesia, including ambulatory surgeries. The standard agent used for spinal anesthesia is called bupivacaine. It's safe and effective, but has a major disadvantage. It has a long duration of action (up to 4 hours), witch can prolong unnecessarily the patient's stay in the recovery room and in hospital.

Another local anesthetic available for spinal anesthesia is 2-chloroprocaine. It has been used since many years, but some serious cases of toxicity in the 80's led to an interruption of its utilization. Those cases have been proven to be associated with the preservative agent (bisulfite) that was added and to the low pH (<3) of the drug.

Since then, 2-chloroprocaine exists in a preservative-free formulation and has been used in thousands of patients worldwide, without any problem. The major advantage of 2-chloroprocaine is its shorter duration of action, permitting a faster recovery from anesthesia, and also permitting a faster discharge from hospital (in a context of ambulatory surgery)

The purpose of this study is to compare the efficacity and the readiness for discharge (from the recovery room, and from hospital) between two local anesthetics, bupivacaine and 2-chloroprocaine, used for spinal anesthesia in elective ambulatory surgeries.

Patients, after consenting for the study, will be randomly assigned to the following groups:

* spinal anesthesia with chloroprocaine 2% 40 mg (2 mL)
* spinal anesthesia with bupivacaine 0,75% 7,5 mg (1 mL)

An "executant anesthesiologist" will be responsible for performing the spinal anesthesia, with a 25 gauge Sprotte needle, at the level L2L3, L3L4 or L4L5. The "responsible anesthesiologist" will only take charge of the patient after the technique, so he stays double-blinded to the local anesthetic used. During surgery, if the patient feels pain, he may receive iv fentanyl, 25-100 µg at every 5 minutes.

Measures will start immediately after the spinal block:

Evaluation of the sensory block height (with ice):

* Every 3 minutes for 15 minutes (time to obtain a block a about T10)
* Every 5 minutes for 45 minutes (surgery)
* Every 10 minutes for 60 minutes, then every 15 minutes until the block regresses to S2 (recovery room and ambulatory surgery unit)

Evaluation of the motor block (using the Bromage scale):

* Every 3 minutes for 15 minutes
* At the beginning and at the end of the surgery
* After the surgery:every 10 minutes for 60 minutes, then every 15 minutes until the block regresses to S2 (recovery room and ambulatory surgery unit)

(Bromage scale: full flexion of feet and knee = 0; able to move knee and feet, not hip = 1; able to move feet only = 2; unable to move feet or knee = 3)

When the block will have regressed to S2, the patient will be asked to urinate. If he isn't able to urinate, this demand will be repeated every 15 minutes. (not applicable if the patient goes home with a urinary catheter)

In the context of an ambulatory surgery, the patient will go home when he will meet the usual discharge criteria. All patients will receive a phone call from the research team the day after surgery, and 7 days later, to assess their satisfaction towards the analgesia and to inquire about potential complications of the spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years and older
* urologic elective ambulatory procedure. For example:cystoscopy, circumcision,transurethral bladder tumor resection, varicocele and hydrocele surgery
* gynecologic elective ambulatory procedure. For example: hysteroscopy, vulvar ou vaginal biopsy
* general surgery elective ambulatory procedure. For example:inguinal herniorraphy, short ano-rectal procedure

Exclusion Criteria:

* INR > 1,3
* platelet < 75 000
* concomitant drugs: clopidogrel (last dose < 7 days), iv heparin, low molecular weight heparin (last dose < 24 hours)
* neurologic disease: spinal stenosis, symptomatic lumbar herniated disc, multiple sclerosis
* liquid restriction (cardiac or renal insufficiency)
* allergy or intolerance to chloroprocaine, bupivacaine or PABA
* atypical plasma cholinesterase or deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Time to obtain discharge criteria from recovery room | within the first hours (1-2 h) after the surgery

SECONDARY OUTCOMES:
Time to obtain discharge criteria from hospital | within the same day of the surgery
The amount of additional IV analgesia (fentanyl) administered during the intraoperative period | total length of surgery
The amount of iv analgesia (fentanyl and morphine) needed in the recovery room | lenght of stay in the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Denis Roy, MD, Study Director — St-Luc hospital, CHUM, University of Montreal; Luc Massicotte, MD, Study Director — St-Luc Hospital, CHUM, University of Montreal; Marie-Andrée Lacasse, MD, resident, Principal Investigator — St-Luc hospital, CHUM, University of Montreal
Locations (1):
- St-Luc Hospital CHUM, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kouri ME, Kopacz DJ. Spinal 2-chloroprocaine: a comparison with lidocaine in volunteers. Anesth Analg. 2004 Jan;98(1):75-80. doi: 10.1213/01.ANE.0000093228.61443.EE. PMID 14693590
- [Background] Smith KN, Kopacz DJ, McDonald SB. Spinal 2-chloroprocaine: a dose-ranging study and the effect of added epinephrine. Anesth Analg. 2004 Jan;98(1):81-88. doi: 10.1213/01.ANE.0000093361.48458.6E. PMID 14693591
- [Background] Vath JS, Kopacz DJ. Spinal 2-chloroprocaine: the effect of added fentanyl. Anesth Analg. 2004 Jan;98(1):89-94. doi: 10.1213/01.ANE.0000093360.02058.ED. PMID 14693593
- [Background] Warren DT, Kopacz DJ. Spinal 2-chloroprocaine: the effect of added dextrose. Anesth Analg. 2004 Jan;98(1):95-101. doi: 10.1213/01.ANE.0000093362.95618.89. PMID 14693594
- [Background] Kopacz DJ. Spinal 2-chloroprocaine: minimum effective dose. Reg Anesth Pain Med. 2005 Jan-Feb;30(1):36-42. doi: 10.1016/j.rapm.2004.09.008. PMID 15690266
- [Background] Davis BR, Kopacz DJ. Spinal 2-chloroprocaine: the effect of added clonidine. Anesth Analg. 2005 Feb;100(2):559-565. doi: 10.1213/01.ANE.0000143381.30409.62. PMID 15673894
- [Background] Yoos JR, Kopacz DJ. Spinal 2-chloroprocaine: a comparison with small-dose bupivacaine in volunteers. Anesth Analg. 2005 Feb;100(2):566-572. doi: 10.1213/01.ANE.0000143356.17013.A1. PMID 15673895
- [Background] Gonter AF, Kopacz DJ. Spinal 2-chloroprocaine: a comparison with procaine in volunteers. Anesth Analg. 2005 Feb;100(2):573-579. doi: 10.1213/01.ANE.0000143380.36298.4A. PMID 15673896
- [Background] Yoos JR, Kopacz DJ. Spinal 2-chloroprocaine for surgery: an initial 10-month experience. Anesth Analg. 2005 Feb;100(2):553-558. doi: 10.1213/01.ANE.0000130397.38849.4A. PMID 15673893
- [Background] Casati A, Danelli G, Berti M, Fioro A, Fanelli A, Benassi C, Petronella G, Fanelli G. Intrathecal 2-chloroprocaine for lower limb outpatient surgery: a prospective, randomized, double-blind, clinical evaluation. Anesth Analg. 2006 Jul;103(1):234-8, table of contents. doi: 10.1213/01.ane.0000221441.44387.82. PMID 16790659
- [Background] Casati A, Fanelli G, Danelli G, Berti M, Ghisi D, Brivio M, Putzu M, Barbagallo A. Spinal anesthesia with lidocaine or preservative-free 2-chlorprocaine for outpatient knee arthroscopy: a prospective, randomized, double-blind comparison. Anesth Analg. 2007 Apr;104(4):959-64. doi: 10.1213/01.ane.0000258766.73612.d8. PMID 17377114
- [Derived] Lacasse MA, Roy JD, Forget J, Vandenbroucke F, Seal RF, Beaulieu D, McCormack M, Massicotte L. Comparison of bupivacaine and 2-chloroprocaine for spinal anesthesia for outpatient surgery: a double-blind randomized trial. Can J Anaesth. 2011 Apr;58(4):384-91. doi: 10.1007/s12630-010-9450-x. Epub 2011 Jan 4. PMID 21203878